CLINICAL TRIAL: NCT04568278
Title: Effect of a Mobile Application System Using the Patient Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) to Improve Patients' Participation in Symptom Management During Cancer Treatment.
Brief Title: Mobile Application Using the PRO-CTCAE to Improve Patients' Participation in Symptom Management During Treatment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Juhee Cho, Director, Cancer Education Center, Samsung Medical Center, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ePRO-CTCAE_2020
Record Dates: First submitted 2020-09-20; First posted 2020-09-29 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms
Keywords: patient-reported outcome; PRO-CTCAE; mobile application; patient engagement
MeSH Terms: conditions — Neoplasms; Patient Participation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, Single center, Open label
Masking Description: Statistician who will analyze the results of the study will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): a mobile application using the PRO-CTCAE along with usual care
  Interventions: Other: ePRO-CTCAE application
- Controlled Group (No Intervention): Usual care

INTERVENTIONS:
Other: ePRO-CTCAE application — The intervention will be the use of a mobile application for recording symptoms during cancer treatments. Patients in the intervention group will have the mobile application (e-PRO) installed on their smart phones on the first day of cancer treatment (chemotherapy or radiation therapy) and patients will be asked to use the application for 8 weeks. Every week, the application will ask patients to report symptoms they experienced during past 7 days using the pre-specified PRO-CTCAE questions for different types of cancer. Patients also can memo and save photos related symptoms using the application and patients can monitor the progression of the symptoms over time.
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the effect of a mobile application system using the Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) to improve patients' participation in symptom management during cancer treatment. Our hypothesis is that patients who use a mobile application using the PRO-CTCAE will more likely to recognize symptoms due to cancer treatment and report them better to their clinicians than patients who do not use the mobile application.

DETAILED DESCRIPTION:
This is a randomized controlled trial to evaluate the effect of a mobile application system using the Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) to improve patients' participation in symptom management during cancer treatment. Breast, lung, head and neck, esophagus, and gynecologic cancer patients who will begin new lines of chemotherapy or radiation therapy will be randomly assigned into the intervention and control groups (2:1 ratio). The intervention group will have the mobile application installed on their smart phones which they could record symptoms and adverse events due to cancer treatments using the pre-specified PRO-CTCAE questions for different types of cancer. The control group will have usual care. Primary endpoint is patients' participation/engagement of reporting symptoms and it will be evaluated at 8 weeks after the intervention using a questionnaire developed by the research team. Secondary end points are unexpected hospital visits during treatment during 8 weeks after the beginning of the treatment and quality of life at 8 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to have chemotherapy or radiation therapy.
* Patients who own a smartphone (Android) and who can use mobile applications.
* Patients who understand the purpose of this study and agree to participate in the study
* Patients age over 18 years old (no age limit, but if necessary informed consent of the caregivers will be obtained for the patients whose age are over 70 years old)

Exclusion Criteria:

* Patients whose life expectancy is less than 6 months (hospice)
* Patients who would any physical or mental problems that would make them difficult to use the applications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Patients' participation in symptom management | 8 weeks after the intervention
  Patients' participation in reporting and managing symptoms due to cancer treatment will be measured using 7 questions developed by study team. Questions will be asked using 4 Likert scale. Minimum value is 0 and maximum value will be 21. Higher score means better outcome.

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C-30 | 8 weeks after the intervention
  State of well-being evaluated by an individual, including both physical, mental, social, and spiritual areas. This will be measured using relevant items of European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Scores will be calculated by manual (0-100) and higher score means better quality of life.
Unexpected visits | 8 weeks after the intervention
  number of unexpected hospital visits (emergency room visits, unplanned outpatient visits, or unplanned hospitalization) due to symptoms or adverse events due to cancer treatment

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Danbee Kang, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee M, Kang D, Kang E, Kim S, Kim Y, Ahn JS, Park S, Lee YY, Oh D, Noh JM, Cho J. Efficacy of the PRO-CTCAE mobile application for improving patient participation in symptom management during cancer treatment: a randomized controlled trial. Support Care Cancer. 2023 May 6;31(6):321. doi: 10.1007/s00520-023-07779-3. PMID 37148373